CLINICAL TRIAL: NCT03814668
Title: Effect of Probiotic Supplementation on Lactose Maldigestion Induced by Lactose Solution: Randomized, Double-blind, Placebo-controlled, Positive-controlled, Three-way Crossover, Acute Lactose Challenge
Brief Title: Effect of Probiotic Supplementation on Lactose Maldigestion Induced by Lactose Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danisco (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: NH-03978
Record Dates: First submitted 2019-01-20; First posted 2019-01-24 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Lactose Intolerance
MeSH Terms: conditions — Lactose Intolerance | interventions — Probiotics; Lactase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotic powder (Experimental): One sachet of Probiotic powderwill be consumed with 25 g lactose in 250 ml of water in the beginning of a 6-hour challenge at the study visits.
  Interventions: Dietary Supplement: Probiotic
- Lactase (Active Comparator): One sachet of Lactase powder will be consumed with 25 g lactose in 250 ml of water in the beginning of a 6-hour challenge at the study visits.
  Interventions: Dietary Supplement: Lactase
- Placebo (Placebo Comparator): One sachet of placebo powder will be consumed with 25 g lactose in 250 ml of water in the beginning of a 6-hour challenge at the study visits.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Intake of probiotic
  Arms: Probiotic powder
Dietary Supplement: Lactase — Intake of lactase
  Arms: Lactase
Other: Placebo — Intake of placebo
  Arms: Placebo

SUMMARY:
Study objectives:

Primary:

Difference in breath hydrogen concentration (BHC, ppm) in lactase and probiotic groups compared to placebo, measured by the incremental area under curve (iAUC) analysis

Non-inferiority in breath hydrogen concentration (BHC, ppm) of probiotic group compared to lactase group, measured by the incremental area under curve (iAUC) analysis

Secondary:

Breath test

* Breath hydrogen peak value (ppm) in lactase and probiotic groups compared to placebo
* Cumulative breath hydrogen (ppm) in lactase and probiotic groups compared to placebo

Acute gastrointestinal symptoms (severity or presence/absence to be defined on a Likert scale) in lactase and probiotic groups compared to placebo

* Abdominal pain
* Flatulence
* Bloating
* Nausea and vomiting
* Bowel movements and diarrhea (if present, stool consistency to be defined on Bristol stool scale and number of bowel movements to be recorded)

Ancillary:

* Baseline fasting BHC (ppm)
* Breath methane CH4 (ppm)
* Breath carbon dioxide CO2 (ppm)
* Probiotic identification in feces before each lactose challenge by molecular methods
* Gene test to determine lactase deficiency status at screening (following SNP variants to be screened: 13910*C (Europe, Central Asia, commonly used) -22018*G (Europe), -13915*T (Saudi-Arabia, Africa), -14010*G (Africa), -13907*C (Africa))

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary, written, informed consent to participate in the study
2. Agreement to comply with the protocol and study restrictions
3. Healthy females and males of age 25 to 60 years (inclusive)
4. Self-declared, suspected or medically diagnosed lactose intolerance
5. Increase of more than 20 ppm in breath hydrogen within 3 h from the baseline fasting breath hydrogen value
6. Participants who agree to maintain their usual dietary habits throughout the trial period
7. Participants who agree not to consume probiotics, prebiotics, fermented milk, and/or yogurt containing probiotics during the intervention period (Visits 3-5) and two weeks before Visit 3 (2 weeks after screening visit)
8. Females of child-bearing potential who agree to use a medically approved method of birth control
9. Ability of the participant (in the investigator's opinion) to comprehend the full nature and purpose of the study including possible risks and side effects
10. Covered by Health Insurance System and / or in compliance with the recommendations of National Law in force relating to biomedical research

Exclusion Criteria:

1. Gastrointestinal disorder or disease (e.g. Crohn's disease, ulcer, irritable bowel syndrome (IBS), Celiac disease, small intestinal bacterial overgrowth (SIBO), pancreatitis and disorders affecting gastrointestinal motility)
2. Diagnosed type 1 or type 2 diabetes
3. Prior abdominal surgery that, in the opinion of the investigator, may present a risk for the participant or affect study results
4. Ongoing or recent (last 1 month) antibiotic treatment.
5. Use of laxatives or drugs known to affect gut motility 1 month preceding the screening visit and during the study
6. Ongoing or recurrent use of proton pump inhibitors
7. Colonoscopy within 3 months before screening
8. History of recurrent colon cleansing and/or a colon cleansing within 3 months before screening
9. Gastrointestinal infection within 1 month before screening or during the trial
10. Clinically significant underlying systemic illness that may preclude the participant's ability to complete the trial or that may affect the study outcomes (e.g. bowel cancer, prostate cancer, terminal illness)
11. History of diagnosed coronary heart disease/cardiovascular disease or artificial heart valve
12. Any obstructive or restrictive respiratory syndrome/disease that may impact breath test (e.g. asthma or chronic obstructive pulmonary disease (COPD))
13. Regular use of tobacco, snuff, nicotine and e-cigarette, and possible other inhaled products. Light smokers (less than 5 cigarettes per day) who agree not to smoke during the whole duration of the study may be included.
14. Self-declared history of alcohol abuse (for females: >3 drinks on any single day and >7 drinks per week; for males: >4 drinks on any single day and >14 drinks per week)
15. Self-declared use of illicit drugs within 4 weeks preceding the screening visit
16. Pregnant or lactating female, or pregnancy planned during study period
17. Participants under administrative or legal supervision.
18. Participation in another study with any investigational product within 60 days of screening
19. Clinically significant abnormal values in safety blood tests at screening
20. Other reasons that, in the opinion of the Investigator, make the participant unsuitable for enrolment
21. Who would receive more than 4500€ as indemnities for his participation in biomedical research within the last 12 months, including the indemnities for the present study.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Difference in breath hydrogen concentration (BHC, ppm) in probiotic group compared to placebo | During the 6-hour acute lactose challenge
  Difference in breath hydrogen concentration (BHC, ppm) in probiotic compared to placebo, measured by the iAUC analysis
Difference in breath hydrogen concentration (BHC, ppm) in lactase group compared to placebo | During the 6-hour acute lactose challenge
  Difference in breath hydrogen concentration (BHC, ppm) in lactase group compared to placebo, measured by the iAUC analysis
Non-inferiority in breath hydrogen concentration (BHC, ppm) of probiotic group compared to lactase group (positive control) | During the 6-hour acute lactose challenge
  Non-inferiority in breath hydrogen concentration (BHC, ppm) of probiotic group compared to lactase group (positive control), measured by the iAUC analysis

SECONDARY OUTCOMES:
Difference in breath hydrogen concentration (BHC, ppm) in lactase group compared to placebo, measured by breath hydrogen peak value | During the 6-hour acute lactose challenge
  Difference in breath hydrogen concentration (BHC, ppm) in lactase group compared to placebo, measured by breath hydrogen peak value
Difference in breath hydrogen concentration (BHC, ppm) in probiotic group compared to placebo, measured by breath hydrogen peak value | During the 6-hour acute lactose challenge
  Difference in breath hydrogen concentration (BHC, ppm) in probiotic group compared to placebo, measured by breath hydrogen peak value
Difference in breath hydrogen concentration (BHC, ppm) in lactase group compared to placebo, measured by cumulative breath hydrogen value | During the 6-hour acute lactose challenge
  Difference in breath hydrogen concentration (BHC, ppm) in lactase group compared to placebo, measured by cumulative breath hydrogen value
Difference in breath hydrogen concentration (BHC, ppm) in probiotic group compared to placebo, measured by cumulative breath hydrogen value | During the 6-hour acute lactose challenge
  Difference in breath hydrogen concentration (BHC, ppm) in probiotic group compared to placebo, measured by cumulative breath hydrogen value
Difference in the severity of abdominal pain in lactase group compared to placebo, as defined by the gastrointestinal symptom survey | During the 6-hour acute lactose challenge
  Difference in the severity of abdominal pain in lactase group compared to placebo, as defined by the gastrointestinal symptom survey
Difference in the severity of abdominal pain in probiotic group compared to placebo, as defined by the gastrointestinal symptom survey | During the 6-hour acute lactose challenge
  Difference in the severity of abdominal pain in probioticgroup compared to placebo, as defined by the gastrointestinal symptom survey
Difference in the severity of flatulence in lactase group compared to placebo, as defined by the gastrointestinal symptom survey | During the 6-hour acute lactose challenge
  Difference in the severity of flatulence in lactase group compared to placebo, as defined by the gastrointestinal symptom survey
Difference in the severity of flatulence in probiotic group compared to placebo, as defined by the gastrointestinal symptom survey | During the 6-hour acute lactose challenge
  Difference in the severity of flatulence in probiotic group compared to placebo, as defined by the gastrointestinal symptom survey
Difference in the severity of bloating in lactase group compared to placebo, as defined by the gastrointestinal symptom survey | During the 6-hour acute lactose challenge
  Difference in the severity of bloating in lactase group compared to placebo, as defined by the gastrointestinal symptom survey
Difference in the severity of bloating in probiotic group compared to placebo, as defined by the gastrointestinal symptom survey | During the 6-hour acute lactose challenge
  Difference in the severity of bloating in probiotic group compared to placebo, as defined by the gastrointestinal symptom survey
Difference in the severity of nausea in lactase group compared to placebo, as defined by the gastrointestinal symptom survey | During the 6-hour acute lactose challenge
  Difference in the severity of nausea in lactase group compared to placebo, as defined by the gastrointestinal symptom survey
Difference in the severity of nausea in probioticgroup compared to placebo, as defined by the gastrointestinal symptom survey | During the 6-hour acute lactose challenge
  Difference in the severity of nausea in probiotic group compared to placebo, as defined by the gastrointestinal symptom survey
Difference in the presence of vomiting in lactase group compared to placebo, as defined by the gastrointestinal symptom survey | During the 6-hour acute lactose challenge
  Difference in the presence of vomiting in lactase group compared to placebo, as defined by the gastrointestinal symptom survey
Difference in the presence of vomiting in probiotic group compared to placebo, as defined by the gastrointestinal symptom survey | During the 6-hour acute lactose challenge
  Difference in the presence of vomiting in probiotic group compared to placebo, as defined by the gastrointestinal symptom survey
Difference in the presence of bowel movements in lactase group compared to placebo, as defined by the gastrointestinal symptom survey | During the 6-hour acute lactose challenge
  Difference in the presence of bowel movements in lactase group compared to placebo, as defined by the gastrointestinal symptom survey
Difference in the presence of bowel movements in probiotic group compared to placebo, as defined by the gastrointestinal symptom survey | During the 6-hour acute lactose challenge
  Difference in the presence of bowel movements in probiotic group compared to placebo, as defined by the gastrointestinal symptom survey
Difference in the presence of diarrhea in lactase group compared to placebo, as defined by the gastrointestinal symptom survey | During the 6-hour acute lactose challenge
  Difference in the presence of diarrhea in lactase group compared to placebo, as defined by the gastrointestinal symptom survey
Difference in the presence of diarrhea in probiotic group compared to placebo, as defined by the gastrointestinal symptom survey | During the 6-hour acute lactose challenge
  Difference in the presence of diarrhea in probiotic group compared to placebo, as defined by the gastrointestinal symptom survey

OTHER OUTCOMES:
Difference in baseline fasting BHC (ppm) between the treatments | Baseline
  Difference in baseline fasting BHC (ppm) between the treatments
Difference in breath methane concentration (ppm) between the treatments | During the 6-hour acute lactose challenge
  Difference in breath methane concentration (ppm) between the treatments
Difference in breath carbon dioxide concentration (ppm) between the treatments | During the 6-hour acute lactose challenge
  Difference in breath methane concentration (ppm) between the treatments
Difference in the quantity of probiotic in fecal samples between the treatments | 48-hours before the visits
  Difference in the quantity of probiotic in fecal samples between the treatments
Description of the SNP variants in each treatment group | At screening
  Description of the SNP variants in each treatment group

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofins Optimed, Gières, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rasinkangas P, Forssten SD, Marttinen M, Ibarra A, Bothe G, Junnila J, Uebelhack R, Donazzolo Y, Ouwehand AC. Bifidobacterium animalis subsp. lactis Bi-07 supports lactose digestion in vitro and in randomized, placebo- and lactase-controlled clinical trials. Am J Clin Nutr. 2022 Dec 19;116(6):1580-1594. doi: 10.1093/ajcn/nqac264. PMID 36149331